CLINICAL TRIAL: NCT03934073
Title: Evaluation of the Benefit of the Training of the Manual Dexterity Post-stroke: Effect on the Function and Spontaneous Use of the Hand and the Cerebral Plasticity
Brief Title: Evaluation of the Benefit of the Training of the Manual Dexterity Post Stroke.
Acronym: DEXTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Centre Hospitalier Sainte Anne
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Vascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DEXTRAIN (Experimental): The DexTrain group sessions will consist of 20 minutes of conventional training followed by 40 minutes of exercises using the DexTrain targeting dexterity components.
  Interventions: Other: DEXTRAIN
- CONVENTIONNELLE (Active Comparator): Conventional training involving stretching of the spastic muscles as well as a set of exercises conventionally used in the protocols of post-stroke rehabilitation (repeated movements, manipulation of objects).
  Interventions: Other: CONVENTIONNELLE
- CONTROLE (Other): To compare the results of SMT and functional MRI.
  Interventions: Other: CONTROLE

INTERVENTIONS:
Other: DEXTRAIN — 12 sessions of 1 hour of rehabilitation (3 sessions / 4 weeks) for the DexTrain group will consist of 20 minutes of conventional training followed by 40 minutes of exercises using the DexTrain targeting the dexterity components.
  Arms: DEXTRAIN
Other: CONVENTIONNELLE — 12 sessions of 1 hour of rehabilitation (3 sessions / 4 weeks) Conventional will be constituted of conventional training consisting of stretching of the spastic muscles as well as exercises used classically in the protocols of rehabilitation post-stroke
  Arms: CONVENTIONNELLE
Other: CONTROLE — Only one assessment will be provided for the control group which will include, Box & Blocks Test (BBT), FFM Dexterity Assessment, Moberg Pick-Up Test (MPUT), Maximal Finger Tapping Rate, Proprioception, SMT, fMRI, Spontaneous hand activity (accelerometry / portable electromyography)
  Arms: CONTROLE

SUMMARY:
Stroke is the second leading cause of death and disability in France: more than half of stroke survivors have a disabling motor deficit, affecting mainly the upper limb. A lack of hand control makes everyday tasks more difficult and reduces the quality of life. The investigators lack approaches to specifically rehabilitate the hand after stroke.

Recently, a new tool has been developed to measure manual dexterity (the Finger Force Manipulandum or FFM). This tool, which records the forces applied by the fingers on pistons, allows to measure more finely the key components of manual dexterity during visuomotor tasks. The tool measures the ability to control and release the force applied by the fingers, to perform sequences, to track and maintain a frequency of tapping (temporality of movement) with the fingers, and to use the fingers independently one another.

DETAILED DESCRIPTION:
The DexTrain proof-of-concept study aims to evaluate the benefit of a training using a tool, an improved version of the FFM, named DexTrain, for the rehabilitation and specific training of the fingers in subjects suffering from stroke. In this study the investigators will compare the effect of conventional therapy with that of the DexTrain method, particularly on the function of the hand and its spontaneous use at home (ecological condition). To better understand the mechanisms involved, the investigators will also study brain plasticity using Transcranial Magnetic Stimulation (SMT) and Functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

Patient :

* At least 18 years old
* 1st symptomatic stroke, due to acute vascular injury (ischemic or haemorrhagic) affecting a single arterial territory dating from 3 months or more (multiple territory: corresponds to a bi-hemispheric or vertebrobasilar stroke and carotid for ischemic and bi-hemispherical stroke for hemorrhagic stroke)
* With a slight-to-moderate deficit of manual dexterity, indicated by a difficulty in picking up blocks in the Box and Block test (<52 blocks / minute, minimum 1 block) as well as an expansion capacity of 10 ° wrist and metacarpophalangeal joints of the index and middle finger.
* Affiliated to a social security scheme, Universal Health Cover or any other equivalent plan.

Volunteers :

* At least 18 years old
* Healthy subject of any disease affecting the hand,

Exclusion Criteria:

* Significant disability or pre-existing deficiency that may interfere with study-specific assessments:

  • History of symptomatic stroke
* Disorders of the understanding not allowing a good comprehension of the tests of motor skills (severe aphasia, dementia, etc.) evaluated by the MMSE (<25)
* Botulinum toxin treatment of spastic muscles of the upper limb less than three months before inclusion and / or during rehabilitation (4 weeks).
* Another severe disease making follow-up difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Change of Box and Block test score | one month
  Change of the Box and Block test score, a measure of the number of blocks the subject can move in 1min, between the beginning (T0) and immediately after the end of treatment (T1). Range of score 0-120. A positive change represents improved performance on Box and Blocks test.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis MAS, PUPH, Principal Investigator — Centre Hospitalier Sainte Anne
Locations (1):
- GHU Paris-Psychiatrie & Neurosciences, Paris, France

REFERENCES:
- [Derived] van Ravestyn C, Gerardin E, Teremetz M, Hamdoun S, Baron JC, Calvet D, Vandermeeren Y, Turc G, Maier MA, Rosso C, Mas JL, Dupin L, Lindberg PG. Post-Stroke Impairments of Manual Dexterity and Finger Proprioception: Their Contribution to Upper Limb Activity Capacity. Neurorehabil Neural Repair. 2024 May;38(5):373-385. doi: 10.1177/15459683241245416. Epub 2024 Apr 4. PMID 38572686
- [Derived] Teremetz M, Hamdoun S, Colle F, Gerardin E, Desvilles C, Carment L, Charron S, Cuenca M, Calvet D, Baron JC, Turc G, Maier MA, Rosso C, Mas JL, Lindberg PG. Efficacy of interactive manual dexterity training after stroke: a pilot single-blinded randomized controlled trial. J Neuroeng Rehabil. 2023 Jul 18;20(1):93. doi: 10.1186/s12984-023-01213-9. PMID 37464404